CLINICAL TRIAL: NCT01818817
Title: Single Injection, Ultrasound Guided Paravertebral Block for Anesthesia in Breast Surgery.
Brief Title: Ultrasound Paravertebral Block in Breast Surgery.
Status: Completed | Type: Observational
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Massimiliano Carassiti, MD, Campus Bio-Medico University
Other Study IDs: CarGal2; TPVB (Other: CampusBioMedico)
Record Dates: First submitted 2013-03-23; First posted 2013-03-27 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2011-09

CONDITIONS: Breast Cancer
Keywords: Ultrasound-guided paravertebral block; regional anesthesia; breast surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- TPVB group: In this group of patients thoracic paravertebral block is performed.
- GA group: In this group of patients general anesthesia is performed.

SUMMARY:
The purpouse of the study is to determine wether Ultrasound Guided,Ens-assisted paravertebral block with single shot is a safe and reliable anesthetic technique in breast surgery.

DETAILED DESCRIPTION:
General anaesthesia is currently the conventional technique used for breast surgery. Thoracic Paravertebral block (PVB) has been used with multiple injection.

We compared a single injection thoracic PVB with general anaesthesia (GA) in 20 consenting patients, scheduled for unilateral breast surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists classification I-III
* Written informed consent
* Age older than 18 years old

Exclusion Criteria:

* allergy to local anesthetics
* local sepsis

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient candidate for minor breast surgery.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | Up to 24 hours
  The anesthesist evaluated the post-operative pain at rest and in movement with the NRS at 3-6-12-24 hours.

SECONDARY OUTCOMES:
Consumption of analgesic drugs | up to 24 hours
  We register the consumption of analgesic drugs in both groups in the post-operative period till 24 hours.
Efficacy of Paravertebral block | pre-operative
  We evaluate efficacy and extension of the block with ice test and pin-prick test

OTHER OUTCOMES:
Post-operative nausea and vomit | up to 24 hours
  We register the incidence of nausea and vomit in the post-perative time.
Appreciation of patients | At 24 hours
  We administer an assessment questionnaire to patients to evaluate the appreciation of the anesthesiologic technique

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano Carassiti, MD, Principal Investigator — Campus Bio Medico
Locations (1):
- Campus Bio Medico, Rome, RM, Italy